CLINICAL TRIAL: NCT05985538
Title: Impact of E-Cigarette Prevention Messages on Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-1245; 5R01DA049155-02 (NIH)
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Vaping Behavior
Keywords: Health communication; Tobacco use; vaping prevention
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaping prevention text messages (Experimental): Participants will receive text messages (2 daily, on average) about the harms of e-cigarette use and vaping for 28 days, with introductory messages sent on day 1 and concluding messages sent on day 28.
  Interventions: Behavioral: Vaping prevention text messages
- Wellness behavior text messages (Active Comparator): Participants will receive text messages (2 daily, on average) about general wellness topics, with introductory messages sent on day 1 and concluding messages sent on day 28.
  Interventions: Behavioral: Wellness behaviors text messages

INTERVENTIONS:
Behavioral: Vaping prevention text messages — Participants will receive text messages (2 daily, on average) about the harms of e-cigarette use and vaping for 28 days, with introductory messages sent on day 1 and concluding messages sent on day 28. Each vaping prevention text message will focus on one of six topics: nicotine addiction, monetary costs of vaping, chemical exposures from e-cigarette vapor, cosmetic effects of vaping, mental and physical use symptoms of vaping, and health impact on organs from vaping. Some text messages will ask participants for a reply (i.e., two-way messages).
  Arms: Vaping prevention text messages
Behavioral: Wellness behaviors text messages — Participants will receive text messages (2 daily, on average) about general wellness topics, with introductory messages sent on day 1 and concluding messages sent on day 28. Each wellness text message will focus on one of six topics: sleep hygiene, safe driving, sun safety, study habits, nutrition, and exercise. This attention control condition is matched with the intervention condition in that participants will receive the same number of text messages over the same number of days, the same intervention structure (e.g., 6 topics), and the same number and types of two-way messages.
  Arms: Wellness behavior text messages

SUMMARY:
The purpose of this trial is to determine whether a vaping prevention text message program reduces susceptibility to vaping among adolescents and young adults. This study addresses this issue by exposing participants to a vaping prevention text message program over a 28-day period in a randomized controlled trial with a matched attention control condition. A follow-up assessment is also made 4 weeks after the text messaging ends.

DETAILED DESCRIPTION:
Tobacco prevention communication is a key tool for reducing tobacco use among adolescents and young adults. While the use of e-cigarettes and vaping has increased greatly among adolescents and young adults, there has been a dearth of research on effective communication strategies to reduce vaping. This study will test the impact of a text-messaging program on reducing susceptibility to vaping in a randomized controlled trial, illuminating whether such programs can be effective. The investigators focus on adolescents and young adults (ages 13-20) who currently vape or who are at risk of vaping.

Participants will be randomly assigned to receive either a vaping prevention text message program or a wellness text message program (control). Participants in the study will take 4 online surveys over an 8-week period - at Visit 1 (baseline), Visit 2 (2 weeks), Visit 3 (4 weeks), and Visit 4 (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-20 years old (inclusive)
* Have a phone that sends and receives text messages
* Ever vaped or are susceptible to using e-cigarettes or vaping

Exclusion Criteria:

* None

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 480 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Noar, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Started | 239 | 241
Completed | 180 | 177
Not Completed | 59 | 64

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages | Total
Number analyzed (Participants) | 239 | 241 | 480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 161 | 133 | 294
  Between 18 and 65 years | 78 | 108 | 186
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.59 (1.75) | 17.76 (1.99) | 17.68 (1.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The following data excludes participants who did not select male or female.
  Participants
    number analyzed (Participants) | 229 | 225 | 454
    Female | 130 | 123 | 253
    Male | 99 | 102 | 201
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 44 | 95
  White | 146 | 149 | 295
  More than one race | 20 | 23 | 43
  Unknown or Not Reported | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  United States | 239 | 241 | 480
Mean Susceptibility to Vaping Score [Mean (Standard Deviation); unit: units on a scale] — The mean susceptibility to vaping score will be assessed using the questionnaire. Response options are on a 1 to 4 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-4), with higher scores representing a greater susceptibility to vaping (a worse outcome).
  units on a scale | 2.10 (.96) | 2.13 (.89) | 2.11 (.92)

OUTCOME MEASURES:

1. Primary Outcome: Mean Susceptibility to Vaping Score
Description: The mean susceptibility to vaping score will be assessed using the questionnaire. Response options are on a 1 to 4 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-4), with higher scores representing a greater susceptibility to vaping (a worse outcome).
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 1.91 (1.01) | 1.82 (0.88)

2. Secondary Outcome: Mean Vaping Instrumental Attitudes Score
Description: The mean vaping instrumental attitudes score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores representing a belief that vaping is more beneficial, safe and healthy.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 1.56 (0.82) | 1.67 (0.79)

3. Secondary Outcome: Mean Vaping Affective Attitudes Score
Description: .The mean vaping affective attitudes score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores representing a belief that vaping is more enjoyable, pleasant, and fun.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 2.31 (1.13) | 2.28 (1.16)

4. Secondary Outcome: Mean Vaping Addiction Risk Beliefs Score
Description: The mean vaping addiction risk beliefs score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores representing more tendency to addiction.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 3.70 (1.30) | 3.28 (1.29)

5. Secondary Outcome: Mean Vaping Monetary Cost Beliefs Score
Description: The mean vaping monetary cost beliefs score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores represents participants' believes that vaping is a costly activity.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 3.63 (1.50) | 3.46 (1.51)

6. Secondary Outcome: Mean Vaping Chemical Risk Beliefs Score
Description: The mean vaping chemical risk beliefs score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores representing participant's believes that e-cigarette vapor contains chemicals that pose health risks.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 4.16 (1.09) | 4.04 (1.19)

7. Secondary Outcome: Mean Vaping Cosmetic Risk Beliefs Score
Description: The mean vaping cosmetic risk beliefs score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores representing participant belief that use will harm their cosmetic appearance.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 3.97 (1.09) | 3.63 (1.25)

8. Secondary Outcome: Mean Vaping Health Symptoms Beliefs Score
Description: The mean vaping physical symptoms of use beliefs score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores represent participant believes that e-cigarette use will cause certain physical symptoms.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 3.92 (1.09) | 3.77 (1.15)

9. Secondary Outcome: Mean Vaping Mental Health Symptoms of Use Beliefs Score
Description: The mean vaping mental health symptoms of use beliefs score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores represent participant believes that e-cigarette use will cause or worsen mental health symptoms.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 3.82 (1.13) | 3.39 (1.23)

10. Secondary Outcome: Mean Vaping Health Organ Risk Beliefs Score
Description: The mean vaping health organ risk beliefs score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores representing participant believes that e-cigarette use will harm the health of certain organs.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 4.19 (1.04) | 4.02 (1.13)

11. Secondary Outcome: Mean Susceptibility to Smoking Cigarettes Score
Description: The mean susceptibility to smoking cigarettes score will be assessed using the questionnaire. Response options are on a 1 to 5 scale. Overall scale scores are determined by summing scores of the 3 items and dividing them by 3 (range 1-5), with higher scores represent participant more open to smoking.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 1.46 (.78) | 1.42 (.70)

12. Secondary Outcome: Mean Smoking Instrumental Attitude Score
Description: The 1-item mean smoking instrumental attitude measure assesses a participant's attitude toward smoking. Response options are on a 1 to 5 scale, with higher scores representing a more harmful perception of smoking.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 1.41 (.85) | 1.39 (.87)

13. Secondary Outcome: Mean Smoking Affective Attitude Score
Description: The 1-item mean smoking affective attitude measure assesses a participant's attitude toward smoking (unenjoyable/enjoyable). Response options are on a 1 to 5 scale, with higher scores representing a more enjoyable attitude toward smoking.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 2.01 (1.24) | 1.85 (1.14)

14. Secondary Outcome: Mean Smoking Addiction Risk Belief Score
Description: The 1-item mean smoking addiction risk belief measure assesses the extent to which a participant believes that smoking will lead to addiction. Response options are on a 1 to 5 scale, with higher scores representing beliefs that smoking will lead to addiction.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 3.98 (1.41) | 4.04 (1.37)

15. Secondary Outcome: Mean Smoking Health Harm Risk Belief Score
Description: The 1-item mean smoking health harm risk belief measure assesses the extent to which a participant believes that smoking will lead to health harm. Response options are on a 1 to 5 scale, with higher scores representing higher beliefs that smoking will cause to health harm.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 4.25 (1.25) | 4.28 (1.26)

16. Secondary Outcome: Mean Vaping Injunctive Norms Score
Description: The 3-item mean vaping injunctive norms scale assesses a participant's perception of others' approval or disapproval of their vaping behavior. Response options are on a 1 to 5 scale. Overall scores are determined by summing the scores of the 3 items and dividing them by 3 (range 1-5), with higher scores representing a participant's perception of others' approval about vaping.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 4.37 (.88) | 4.31 (1.07)

17. Secondary Outcome: Mean Vaping Refusal Self-efficacy Score
Description: The 3-item mean vaping refusal self-efficacy scale assesses a participant's confidence that they could refuse to vape in a social situation. Response options are on a 1 to 5 scale. Overall scores are determined by summing the scores of the 3 items and dividing them by 3 (range 1-5), with higher scores representing a higher amount of refuse to vape in a social situation.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
score on a scale | 3.86 (1.25) | 3.90 (1.24)

18. Secondary Outcome: Frequency of Vaping
Description: Participants will be asked the number of days they vaped over the past 30 days, with higher scores indicating more days vaped.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
days | 5.54 (14.84) | 5.80 (16.87)

19. Secondary Outcome: Frequency of Cigarette Smoking
Description: Participants will be asked the number of days they smoked cigarettes over the past 30 days, with higher scores indicating more days smoked.
Time Frame: Visit 3 (4 weeks)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
days | 4.02 (16.86) | 4.23 (17.58)

20. Secondary Outcome: Frequency of Using Other Tobacco Products
Description: Participants will be asked if they used other tobacco products (OTP) over the past 30 days. OTP use will be determined as follows: no use = person who doesn't use OTPs; used = person who uses OTPs; no response = person who skipped or refused to answer
Time Frame: Visit 3 (4 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
Number analyzed (Participants) | 239 | 241
Participants
  No use | 71 | 83
  Used | 160 | 152
  No response | 8 | 6

ADVERSE EVENTS:
Description: The protocol does not require Adverse Event Collections and/or All-Cause Mortality data. Adverse Events were not monitored/assessed. Therefore, the total Number of Participants at Risk (e.g., "All-Cause Mortality, Serious, and Other [Not Including Serious] was entered as "0".
Arm/Group | Vaping Prevention Text Messages | Wellness Behavior Text Messages
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05985538/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05985538/SAP_001.pdf